CLINICAL TRIAL: NCT02801383
Title: Randomized, Double-blind, Parallel, Controlled Clinical Study to Evaluated the Efficacy and Safety of Recombinant Human Interferon Alpha-2b Gel (Yallaferon®) in HPV-16 and/or HPV-18 Infection
Brief Title: Recombinant Human Interferon a-2b Gel for HPV-16 and/ or HPV-18 Gynecological Infections
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lee's Pharmaceutical Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Zhaoke-201509-RHI
Record Dates: First submitted 2016-06-12; First posted 2016-06-15 (Estimated); Last update posted 2016-06-15 (Estimated); Status verified 2016-06

CONDITIONS: Cervical HPV-16 and / or HPV-18 Infection
MeSH Terms: interventions — Gels

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Treatment group (Active Comparator): received 1g recombinant human α-2b interferon gel every other day for consecutive 6-10 courses of treatment
  Interventions: Drug: Yallaferon®， the recombinant human interferon α-2b gel
- controlled group (Placebo Comparator): received 1g gel (without biological active ingredient) every other day for consecutive 6-10 courses of treatment
  Interventions: Other: gel without active ingredient

INTERVENTIONS:
Drug: Yallaferon®， the recombinant human interferon α-2b gel
  Arms: Treatment group
Other: gel without active ingredient
  Arms: controlled group

SUMMARY:
to assess the efficacy and safety of recombinant human interferon α-2b gel (Yallaferon®) for the treatment of patients with cervical HPV-16 and/or HPV-18 infections; to analyze the HPV type infections and clinical negative conversion.

DETAILED DESCRIPTION:
100 patients with positive HPV-16 and HPV-18 infection are randomized into interferon gel group and control group at ratio of 1:1 (50 patients in treatment group and 50 patients in control group). The patients in treatment group received 1g recombinant human α-2b interferon gel every other day for consecutive 6-10 courses of treatment, whereas no treatment was conducted in control group.

ELIGIBILITY:
Inclusion Criteria:

* Age 25 to 65 years of age with the sex life of female patients;
* HPV DNA typing test for HPV-16 and/ or HPV-18 positive in 1 month.

Exclusion Criteria:

* Patients with cervical intraepithelial neoplasia Ⅱ / Ⅲ, cervical cancer;
* Associated with fungal vaginitis, trichomonas vaginitis, HIV positive patients;
* Associated with acute, severe bacterial or viral infection;
* Autoimmune diseases;
* Within 3 months before screening patients used corticosteroids, immunosuppressants or other antiviral drugs;
* Allergies or allergy to the drug known ingredients;
* History of suffering CNS diseases, epilepsy and/or psychological disorder;
* Pregnant and lactating women;
* The researchers do not consider it appropriate clinical trials.

Ages: 25 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-09; Primary Completion 2017-03 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
difference of HPV-16 and/ or HPV-18 DNA negative conversion rate | three months
  Primary efficacy endpoint was the difference of HPV-16 and/ or HPV-18 DNA negative conversion rate on the 3th month between the two groups.

SECONDARY OUTCOMES:
difference of HPV-16 and/ or HPV-18 DNA negative conversion rate | six months, nine months and twelve months
  Secondary efficacy endpoint was the difference of HPV-16 and/ or HPV-18 DNA negative conversion rate on the 6th, 9th and 12th month between the two groups.
The recurrent rate of HPV-16 and/ or HPV-18 DNA among patients with negative-conversion result between the two groups | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University First Hospital, Beijing, China